CLINICAL TRIAL: NCT06474130
Title: Cervical Sensorimotor Control Assessment Using a Virtual Reality System in Individuals With and Without Chronic Neck Pain
Brief Title: Assessing Cervical Sensorimotor Control With VR in Chronic Neck Pain
Status: Recruiting | Type: Observational
Sponsor: National Cheng Kung University (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, YI-JU TSAI, professor, National Cheng Kung University
Other Study IDs: NCKU_VR
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Neck Pain; Virtual Reality; Sensorimotor
Keywords: Sensorimotor control; Virtual Reality; Chronic neck Pain; cervical
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic neck pain group: Pain was unilateral or bilateral between the superior nuchal line and 1st thoracic vertebra; Neck pain persisting for 3 months and above; Average pain intensity of last pain episode was between 2 and 8 based on the numerical rating scale (NRS).
- Healthy adults group: Do not have any complaints of current pain and impairments of neuromusculoskeletal systems within the last 6 months.

SUMMARY:
To develop a cervical SMC VR assessment system incorporating different SMC tests and to compare cervical SMC performance using this self-developed VR assessment system in individuals with and without CNP

ELIGIBILITY:
Inclusion Criteria:

1. For patients with chronic neck pain:

   * Pain was unilateral or bilateral between the superior nuchal line and 1st thoracic vertebra,
   * Neck pain persisting for 3 months and above,
   * Average pain intensity of last pain episode was between 2 and 8 based on the numerical rating scale (NRS)
2. Healthy asymptomatic adults:

   * Do not have any complaints of current pain and impairments of neuromusculoskeletal systems within the last 6 months

Exclusion Criteria:

* acute or the first onset of neck pain
* previous fracture or surgery of the spine
* diagnosed cardiopulmonary diseases, for example, chronic obstructive pulmonary disease, pulmonary tuberculosis, asthma, chronic bronchitis, pulmonary emphysema
* diagnosed gastrointestinal and abdominal conditions which may interfere daily activities within the past 6 months
* medical conditions that may affect balance and study procedures (e.g. neurological diseases, vestibular disorders, malignant tumors)
* metabolic diseases such as anemia and diabetes
* smoking, plan to pregnant or in pregnancy
* psychological disorders (affect questionnaire responses)
* unable to walk independently
* Corrected visual abnormalities or individuals unable to wear contact lenses for vision correction due to the potential interference of wearing VR head-mounted display with glasses

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with CNP will be recruited from the affiliated hospital, local outpatient clinics, local communities and around the campus.
  Healthy adults will be recruited from the local communities near the university in the Tainan city.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Cervical Range of Motion (ROM) | One day
  Participants will follow the instructions that appeared in the VR HMD to perform active maximal neck flexion, extension, side bending and rotation. The maximal ROM in each direction will be calculated and obtained based on the IMU sensors embedded in the HMD.
Joint Position Error (JPE) | One day
  There will be a virtual target displayed in the VR HMD. Participant will be instructed to remember this position, then close their eyes and move the head away from the target center, and then return to the initial starting position.
  Difference between the starting position and final position in distance (mm) will be calculated.
Figure of Eight (FOE) | One day
  The participant will be instructed to control the red dot moving along the path of the figure-of-eight as accurately as possible by moving their head.
Subjective Visual Vertical (SVV) | One day
  A tilted white rod will be presented at different angles for 1-degree interval from 45 to 135 degrees randomly on the display as described above. The rod will be precisely controlled by using left and right arrow keys of a keyboard. Participants will be instructed to reposition the white rod so that the white rod will be positioned vertically while keeping the head and neck as still as possible.
Head Tile Response (HTR) | One day
  A tilted white rod will be presented at different angles for 1-degree interval from 45 to 135 degrees randomly on the display as described above. Participants will be instructed to tilt their heads laterally so that the line will be re-positioned vertically.
Saccades | One day
  Two virtual white targets at 90 degrees of visual angle positioned 0.82 m apart from the participant will be displayed in the VR HMD. Participants will be asked to shift their gaze quickly between two targets without moving their heads for 10 secs.
Smooth Pursuit Neck Torsion (SPNT) | One day
  A virtual red-dot target is displayed in the VR HMD. The target will move in a horizontal plane with a sinusoidal pattern (30 degrees per second) from left to right and back 10 times with a visual angle of 40 degrees. Participants will be requested to follow the moving target with their eyes and keep their heads still.
Postural Sway (PS) | One day
  Participants will be asked to follow the instructions that appeared in the VR HMD and stand still for 30 seconds in EO or EC condition and in neck neutral or neck torsion 45-degree position

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No